CLINICAL TRIAL: NCT02794090
Title: Exclusive Telephone Coaching in Maintaining Weight Loss - An Randomized Controlled Trial of Childhood Obesity Treatment
Brief Title: Childhood Obesity Treatment - Telephone Coaching vc Usual Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sodertalje Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Pernilla Danielsson, PhD pediatric nurse, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: So100
Record Dates: First submitted 2016-05-31; First posted 2016-06-08 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Childhood Obesity
Keywords: Behavioral treatment; Telephone coaching; Outpatient clinic
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care, individual visits (Active Comparator): Usual care according to regular treatment routines at the clinic during 18 months. The Child and parent(s) at regular visits to the nurse at the clinic.
  Interventions: Behavioral: Usual care, individual visits
- Telephone coaching (Active Comparator): Intervention: Telephone consultation each months except for summer holidays during 18 months. The treating nurse communicated with one of the parents.
  Interventions: Behavioral: Telephone coaching

INTERVENTIONS:
Behavioral: Usual care, individual visits — Randomized controlled study of two types of delivering behavioral treatment to Children suffering from obesity.
  Arms: Usual care, individual visits
Behavioral: Telephone coaching — Randomized controlled study of two types of delivering behavioral treatment to Children suffering from obesity.
  Arms: Telephone coaching

SUMMARY:
This study evaluates if usual physical care visits to an outpatient pediatric clinic can be replaced with more frequent and shorter Telephone coaching Contacts during 18 months.

DETAILED DESCRIPTION:
In this randomized controlled study, patients at age 5 to 14 and enrolled in obesity treatment, were randomized to either usual care according to regular routine or to telephone consultation.The randomization was done at the start of individual treatment and lasted for 18 months. We also studied working time required for the Health care, and the families' experience of the Telephone coaching.

ELIGIBILITY:
Inclusion Criteria:

* Children 5 to 14 years old who were patients at the outpatient pediatric centre
* All families after that the parents had attended at least 4 of 7 meetings in a parental/education group.

Exclusion Criteria:

* Obesity related syndromes
* Non-Swedish speaking families

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2007-05; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in BMI Standard Deviation Score (units) | From start of treatment, during intervention and follow-up. In total mean 3,7 years
  BMI Standard Deviation Score units using the Swedish reference by Karlberg et al 2001.

SECONDARY OUTCOMES:
Working time required for the Health care personnel | During the intervention 18 months
  Mean time for each group measured in minutes
Families experience of the treatment | During the intervention 18 months
  Experience for both the Telephone consultation and usual care by not validated anonymous questionnaires constructed by the researchers in this project

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Danielsson, PhD, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No